CLINICAL TRIAL: NCT01122602
Title: A Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled Trial Assessing the Analgesic Efficacy of a Single, Oral Dose of a Fast Release Aspirin 650 mg in Postsurgical Dental Pain
Brief Title: Evaluate Analgesic Efficacy of Fast Release Aspirin
Acronym: TAROT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15082; 2014-005278-12 (EudraCT Number)
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Drugs, Investigational
Keywords: Aspirin
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicyclic acid (Fast acting Aspirin, BAY1019036)
- Arm 2 (Active Comparator)
  Interventions: Drug: Acetylsalicyclic acid (Aspirin, BAYE4465)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicyclic acid (Fast acting Aspirin, BAY1019036) — Single dose of fast acting aspirin 2 x 325 mg = 650 mg total
  Arms: Arm 1
Drug: Acetylsalicyclic acid (Aspirin, BAYE4465) — Single dose of regular aspirin 2 x 325 mg = 650 mg total
  Arms: Arm 2
Drug: Placebo — Two placebo tablets
  Arms: Arm 3

SUMMARY:
The objective of the study is to evaluate the analgesic efficacy of a single, oral dose of fast release aspirin tablets, 650 mg (2 x 325 mg) compared to regular aspirin tablets, 650 mg (2 x 325 mg) and placebo in subjects with postsurgical dental pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers between 16 to 45 years of age
* Scheduled to undergo surgical removal of either two partial bony impactions or one full bony alone or in combination with a partial bony impaction, soft tissue impaction or erupted third molar. Maxillary third molars may be removed regardless of impaction level
* Use of only short-acting local anesthetic (e.g., mepivacaine or lidocaine) preoperatively, with or without vasoconstrictor and nitrous oxide
* No use of any analgesics, NSAIDs (Nonsteroidal Anti-inflammatory Drugs), aspirin, any other pain reliever Over the Counter (OTC) or prescription, or herbal supplements within 5 days of surgery. Oral contraceptives, prophylactic antibiotics, pre-anesthetic medication, anesthesia during the procedure, or other routine medications to treat benign conditions that would not confound the evaluation of the investigational would be acceptable.
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, NuvaRing, Depo-Provera, or double-barrier and have a negative pregnancy test at Screening and prior to surgery. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy
* Provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial, (subjects < 18 years of age must sign a written assent and have parental or guardian consent)

Exclusion Criteria:

* History of hypersensitivity to aspirin, salicylates, other NSAIDs (Nonsteroidal Antiinflammatory Drugs), acetaminophen, opioid analgesics, and similar pharmacological agents or components of the investigational products, including the placebo
* Lactose intolerance or have had hypersensitivity reactions to lactose containing products
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted), chronic sinusitis or nasal structural abnormalities causing greater than 50 percent obstruction (polyposis nasi, marked septal deviation) that can interfere with the conduct of the study in the judgment of the Investigator
* Current or past history of bleeding disorder(s)
* History of gastrointestinal bleeding or perforation, related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Acute illness or local infection prior to surgery that can interfere with the conduct of the study in the judgment of the Investigator
* Females who are pregnant or lactating
* Positive alcohol breathalyzer test and positive urine drug test prior to surgery

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2010-04-29 (Actual); Primary Completion 2010-07-29 (Actual); Study Completion 2010-08-06 (Actual)

PRIMARY OUTCOMES:
Time to First Perceptible Pain Relief (PR) | 0 to 6 hours
Time to First Perceptible Pain Relief Confirmed | 0 to 6 hours

SECONDARY OUTCOMES:
Time to meaningful pain relief | 0 to 6 hours
Pain Intensity at 10, 20, 30, 40, 50, and 60 minutes and at 2, 3, 4, 5, and 6 hours After Dosing | 10, 20, 30, 40, and 50 minutes and at 1, 2, 3, 4, 5, and 6 hours post-dose
Pain Intensity Difference (PID) at 10, 20, 30, 40, 50, and 60 minutes and at 2, 3, 4, 5, and 6 hours After Dosing | 10, 20, 30, 40, 50, and 60 minutes and at 2, 3, 4, 5, and 6 hours post-dose
Pain Relief at 10, 20, 30, 40, 50, and 60 minutes and at 2, 3, 4, 5, and 6 hours After Dosing | 10, 20, 30, 40, 50, and 60 minutes and at 2, 3, 4, 5, and 6 hours post-dose
Summed Pain Intensity Differences (SPID ) from Hour 0 through Hour 2, Hour 4 and Hour 6 | 0 - 6 hours post-dose
Summed Total Pain Relief (TOTPAR ) from Hour 0 through Hour 2, Hour 4 and Hour 6 | 0-6 hours post-dose
Time to First use of Rescue Medication | 0 to 6 hours
Cumulative Percentage of Subjects Taking Rescue Medication | 1, 2, 3, 4, 5, and 6 hours post-dose
Global Assessment of the Investigational Product as a Pain Reliever at 6 hours After Dosing or Immediately Before the First Intake of Rescue Medication | At 6 hours postdose or immediately before first use of rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Austin, Texas
  - Salt Lake City, Utah

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/